CLINICAL TRIAL: NCT00398697
Title: Phase 1 Trial of the Combination of Perifosine and Gemcitabine
Brief Title: Phase I Perifosine and Gemcitabine Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 102
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2007-01

CONDITIONS: Neoplasms
Keywords: perifosine; gemcitabine
MeSH Terms: conditions — Neoplasms | interventions — perifosine; Gemcitabine

INTERVENTIONS:
Drug: Perifosine
Drug: Gemcitabine

SUMMARY:
This is a study of the drug perifosine in combination with Gemcitabine. Perifosine is an oral anti-cancer agent that has been used in more than 140 people, but has not been combined with other drugs before this study. The study is designed to determine the highest dose of perifosine that can be administered to people every day while they are on a Gemcitabine regimen, without severe or prolonged nausea, vomiting and diarrhea. This study starts with patients taking 50 mg/day and goes up to 150 mg/day. After the highest tolerable dose is found, we will add 10 more patients at that dose.

DETAILED DESCRIPTION:
This is a phase 1, open-label trial of perifosine and gemcitabine in patients with malignancies for whom single agent gemcitabine is a reasonable treatment option. All patients will receive gemcitabine at a dose of 1000 mg/m2 on days 1 and 8 of a 21-day cycle. Patients will receive perifosine orally at a dose of 50, 100 or 150 mg per day for the first 14 days of the 21-day cycle. Cohorts of 3 patients will be treated with doses of 50 mg administered either once, twice or three times a day. In this study a maximum tolerated dose (MTD) will be defined as a dose that can be given without grade 3/4 non-hematologic toxicity in more than 1/3 patients. If 2/3 patients in any cohort encounter a grade 3/4 non-hematologic toxicity, an additional 3 patients will be added. If the dose is intolerable for >3/6 patients then the previous level will be declared the MTD. Once an MTD has been determined an additional 10 patients will be added at the MTD to better define the expected toxicities.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically or cytologically confirmed diagnosis of cancer for which treatment with single agent gemcitabine would be an appropriate treatment option
* At least 18 years of age
* Patients may have received no more than two prior chemotherapy regimens
* Patients must have a life expectancy of more than 3 months.
* Patients must have a performance status of 0 to 2 according to the ECOG criteria
* Patients must have normal organ and marrow function as defined in the protocol.
* Patients must have recovered from any acute toxicity related to prior therapy, including surgery or radiotherapy.
* Patients must be able to ingest oral medications.
* Female patients who are pregnant or lactating are ineligible. All females of childbearing potential must have a negative serum pregnancy test within 72 hours of treatment. Men and women of childbearing potential must agree to employ adequate contraception.
* Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients may not be receiving any other investigational agents or devices.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with perifosine. HIV-positive patients not receiving combination anti-retroviral therapy must be approved by the study chair prior to entry.
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment) or New York Heart Assoc. class II-IV congestive heart failure.
* Radiation therapy to > 50% of marrow producing sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19
Dates: Start 2004-08; Study Completion 2006-01

PRIMARY OUTCOMES:
GI Toxicities

SECONDARY OUTCOMES:
Other toxicities
Disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Robert Birch, Ph.D., Study Director — Keryx / AOI Pharmaceuticals, Inc.
Locations (1):
- Johnson City, Tennessee, United States

REFERENCES:
- [Result] Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 24, No 18S (June 20 Supplement), 2006: 13084